CLINICAL TRIAL: NCT02658370
Title: A Prospective Pilot Study to Evaluate an Animated Home-based Physical Exercise Program as a Treatment Option for Patients With Rheumatoid Arthritis
Brief Title: An Animated Home-based Physical Exercise Program as a Treatment Option for Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eugen Feist (Other)
Responsible Party: Sponsor-Investigator, Eugen Feist, MD, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: EA1/189/10
Record Dates: First submitted 2016-01-13; First posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Rheumatoid Arthritis
Keywords: physical exercises; physical therapy; Wii game console; patients perspective
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- animated home-based exercises (Wii-fit) (Experimental): using the Wii game console by Nintendo
  Interventions: Device: animated home-based exercises (Wii-fit); Procedure: conventional home-based exercise program
- conventional home-based exercise program (Active Comparator): by using a compilation with 31 exercises especially for rheumatoid arthritis patients
  Interventions: Device: animated home-based exercises (Wii-fit); Procedure: conventional home-based exercise program

INTERVENTIONS:
Device: animated home-based exercises (Wii-fit)
  Other Names: software Wii-fit plus
Procedure: conventional home-based exercise program

SUMMARY:
The purpose of this pilot study is to investigate feasibility and patients´ assessment using an animated home-based exercise program (Software Wii-fit of the Nintendo Wii game console) for patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the 1987 and 2010 American College of Rheumatology (ACR) criteria for rheumatoid Arthritis
* Disease activity (patients' global assessment, PtGA) < 30 mm under therapy with a biological DMARD according to label

Exclusion Criteria:

* Epilepsy
* Flare of RA
* A previous use of a Wii console for more than 5 hours

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
feasibility of the animated home-based physical exercise program | 12 weeks
  to be assessed by qualitative interview analysis

SECONDARY OUTCOMES:
muscle strenght measurement | 12 weeks
  isometric measurement of 9 muscle groups by using a handheld dynamometer
6-minute walk test | 12 weeks
  standardised walk test (walk course with a minimum of 30 meters in length) on flat ground where patients can choose their own intensity of exercise and are allowed to stop and rest during the test. total walk distance after 6 minutes will be evaluated.
respiratory function test | 12 weeks
  peak expiratory flow taken by a peak flow meter (liter/ Minute)
Health Assessment Questionnaire Disability Indes (HAQ-DI) | 12 weeks
  standardised Patient reported outcome measurement (8 categories regarding disabilities in daily life)
patient's visual analogue scale for pain | 12 weeks
  patients self-reported judgement on a 100 mm scale
patient's visual analogue scale for disease activity | 12 weeks
  patients self-reported judgement on a 100 mm scale
short form 36 questionnaire (SF36) | 12 weeks
  standardised patient reported outcome measurement (11categories regarding quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Eugen Feist, MD, Principal Investigator — Charité Berlin, Department of rheumatology and clinical immunology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zernicke J, Kedor C, Muller A, Burmester GR, Reisshauer A, Feist E. A prospective pilot study to evaluate an animated home-based physical exercise program as a treatment option for patients with rheumatoid arthritis. BMC Musculoskelet Disord. 2016 Aug 18;17(1):351. doi: 10.1186/s12891-016-1208-3. PMID 27538847